CLINICAL TRIAL: NCT06400615
Title: Phase 2 Safety, Efficacy and, Tolerability of Fixed Dose Combination of Aroxybutynin/Atomoxetine (AD109) in Obstructive Sleep Apnea Patients Taking Tirzepatide, Semaglutide or Liraglutide
Brief Title: Study That Tests AD109 in Patients Taking GLP-1 Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APC-APN-201
Record Dates: First submitted 2024-04-12; First posted 2024-05-06 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: OSA
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: A total of approximately 40 participants will be enrolled in the 2 arms:
  20 subjects taking GLP-1+ AD109 20 subjects taking AD109 without any GLP-1 Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Active Comparator): Twenty patients who are taking GLP-1 at time of enrollment will be treated with AD109
  Interventions: Drug: AD109
- Arm 2 (Active Comparator): Twenty patients who are not taking a GLP-1 will be treated with AD109 only
  Interventions: Drug: AD109

INTERVENTIONS:
Drug: AD109 — Oral administration at bedtime

SUMMARY:
Phase 2 Safety, Efficacy and, Tolerability of Fixed Dose Combination of Aroxybutynin/Atomoxetine (AD109) in Obstructive Sleep Apnea Patients Taking Tirzepatide, Semaglutide or Liraglutide

DETAILED DESCRIPTION:
Study APC-APN-201 is an open-label, parallel-arm, 6 weeks study of AD109 in participants with OSA and obesity. One arm consists of patients concomitantly taking tirzepatide, semaglutide or liraglutide, and a second comparator arm consists of patients not taking any GLP drug but who otherwise would meet the criteria for prescribing a GLP-1 (i.e., BMI≥27). Each arm is composed of approximately 20 participants. The participants on GLP-1 must be on a stable maintenance dose that has remained unchanged for at least four weeks prior to enrollment. All study procedures, including open-label dosing of AD109, are the same for both arms; the arms differ only in concomitant GLP-1 use.

ELIGIBILITY:
Inclusion Criteria:

• Age and Sex Between 18-75 years of age at the time of informed consent.

Body Mass Index (BMI) • BMI between 27 and 43 kg/m2 for men, or 45 kg/m2 for women, inclusive.

Obstructive Sleep Apnea (OSA) History and Measures

* Home Sleep Apnea Testing (HSAT) criteria ( Mean Respiratory Event Index (REI4) (Hypopneas defined by 4% oxygen desaturation) of >5 and <45. REI is determined as a mean number collected across 2 nights of testing initiated at Visit 2; ≤ 25% central or mixed apneas (as proportion of total apneas and hypopneas)
* Participants with a history of using devices for OSA treatment, including Continuous Positive Airway Pressure (CPAP), oral or nasal devices, or positional devices, may enroll as long as the devices have not been used for at least 2 weeks prior to first HSAT and are not used during participation in the study.

Weight

* For the subjects in the incretin arm the following criteria must be met (Patients must have an identified prescriber and adhere to drug labelling considerations; A patient's individual dose is stable over the past 4 weeks without intention to increase to decrease dosing based on side effects or efficacy; Willingness to maintain a medication administration diary during the study.
* The following agents and doses are acceptable to meet inclusion criteria: ( Tirzepatide (Mounjaro®, Zepbound®): doses of 2.5mg, 5mg, 7.5mg, 10mg, 12.5mg, 15mg can be given once weekly by subcutaneous injection; Semagultide (Ozempic®, Wegovy®): doses of 0.25mg, 0.5mg, 1mg, 1.7mg, 2.0, or 2.4mg; Liraglutide (Saxenda®) doses of 0.6 mg, 1.2m mg, 1.8 mg, 2.4 mg, 3.0 mg can be given once weekly by subcutaneous injection)

Other doses prescribed by a physician are acceptable if a stable dose is maintained for 4 weeks or more.

Male participants:

• If male and sexually active with female partner(s) of childbearing potential, participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception (see Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information).

Female participants:

• If a woman of childbearing potential (WOCBP), the participant must agree, from Study Day 1 through 1 week after the last dose of study drug, to practice the protocol specified contraception (See Appendix 4: Contraceptive Guidance and Collection of Pregnancy Information). All WOCBP must have negative result of a serum pregnancy test performed at screening ( Females of non-childbearing potential include postmenopausal or permanently sterile.)

Informed Consent

* Participant voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the Screening Visit procedures.
* Participant must be able to understand the nature of the study and must have the opportunity to have any questions answered.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

* Narcolepsy, restless leg syndrome requiring medication, rapid eye movement (REM) sleep behavior disorder
* Current bothersome symptoms of insomnia (difficulty initiating or maintaining sleep, as distinct from unrefreshing sleep or other symptoms attributable to OSA). Participants being treated for insomnia can be enrolled only if the condition is stable and generally controlled.
* Pierre Robin, Treacher Collins, or other craniofacial malformation syndrome, or grade ≥3 tonsillar hypertrophy.
* Clinically significant or medically uncontrolled cardiovascular disease, e.g., ventricular arrhythmia requiring medical or device therapy, unstable atrial fibrillation (including cardioversion, ablation, or change in antiarrhythmic regimen within past 3 months [patients in whom anticoagulation is indicated must be on such treatment for enrollment], or resting heart rate >100), untreated or unstable coronary artery disease (including revascularization within 3 months), cardiac failure, cerebrovascular event or transient ischemic attack or revascularization within 3 months.
* Neuromuscular disorder (e.g., motor neuron disease, muscular dystrophy, or myopathy, myasthenic syndrome); epilepsy; Parkinson, Alzheimer, or other neurodegenerative disease.
* Schizophrenia, schizoaffective disorder, generalized anxiety disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) or International Classification of Disease tenth edition criteria.
* Attempted suicide within 1 year prior to screening, or current suicidal ideation.
* Severe or frequent constipation considered currently bothersome by the patient, or symptomatic gastric motility disorder.
* Current bothersome symptoms of bladder outlet obstruction including difficulty initiating or maintaining urinary flow, straining, or sensation of incomplete bladder emptying; participants being treated with alpha-1 adrenergic antagonist for benign prostatic hypertrophy can be enrolled only if the condition is stable and generally controlled.
* Active substance use disorder as defined in DSM-5, or other substance use that in the investigator's opinion would present an unreasonable risk to the participant, or which would interfere with their participation in the study or confound study interpretation. Positive screen for drugs with abuse liability is an important but not sole determinant of substance use disorder and study eligibility. Participants who use marijuana daily should be excluded.
* A serious illness or infection in the past 30 days as determined by investigator.
* Clinically significant cognitive dysfunction as determined by investigator.
* Narrow angle glaucoma.
* Women who are pregnant or nursing. Prior/Concomitant Therapy
* Participants with prior use of mandibular advancement devices, nasal devices, or sleeping position devices for the treatment of OSA may enroll as long as the devices are not used during participation in the study.
* Participants with history of chronic oxygen therapy are excluded.
* Participants with implanted devices for the treatment of OSA are excluded (e.g., hypoglossal nerve stimulator, or investigational devices).

Prior/Concurrent Clinical Study Experience

• Use of another investigational agent within 30 days or 5 half-lives, whichever is longer, prior to dosing.

Diagnostic Assessments

* Montgomery-Asberg Depression Rating Scale (MADRS) "Suicidal Thoughts question response of thinking of or planning suicide.
* Systolic blood pressure up to 140 mm Hg or diastolic blood pressure up to 90 mm Hg is allowed in participants not currently treated with antihypertensives. If the participant is under the care of a healthcare provider managing blood pressure and on stable (at least 1 month) antihypertensive therapy, systolic blood pressure up to 145/90 is allowed at enrollment. If initial blood pressure (measured in triplicate, use average of final two readings) is above this enrollment threshold, it may be repeated up to a total of 3 times (each in triplicate) to confirm that the reading was not due to measurement technique or transient factors, with selection of the lowest repeated measure. The determination that blood pressure meets enrollment criteria involves the clinical judgment of the investigator interpreting blood pressure readings.
* Unexplained or new identification of hepatic transaminases (AST or ALT) >2X the upper limit of normal (ULN) generally is exclusionary. However, elevation between 2-2.5 may be allowed with prior consent of the sponsor if evidence suggests it is due to nonalcoholic fatty liver disease (NAFLD) or other condition that would not be expected to acutely worsen or require medical intervention during the course of the study.
* Total bilirubin >1.5X ULN (unless confirmed Gilbert syndrome).
* Estimated glomerular filtration rate < 50 ml/min.
* ECG abnormality indicative of clinically significant cardiac disease that may be adversely affected by AD109 Other Exclusions
* Night- or shift-work sleep schedule which causes the major sleep period to be during the day, including on a rotating basis.
* Frequent travel or jet lag is likely to interfere with study procedures or evaluations.
* Employment as a commercial driver or other vehicle operator (includes independent contractors and ride-share services).
* History of sleepiness-related motor vehicle accident (MVA).
* Unwilling to use specified contraception.
* Any condition that in the investigator's opinion would present an unreasonable risk to the participant, including nature or severity of OSA symptoms, or which would interfere with their participation in the study or confound study interpretation.
* Participant considered by the investigator, for any reason, an unsuitable candidate to receive AD109 or unable or unlikely to understand or comply with the dosing schedule or study evaluations.
* Subjects with a history of gastric weight loss surgery (i.e., sleeve gastrectomy, gastric bypass, adjustable gastric banding, biliopancreatic diversion)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Primary Objective (Adverse Events) | 6 weeks
  General safety and tolerability will be assessed between treatment cohorts using the occurrence of spontaneously reported adverse events (AEs) at 6 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Monroe Biomedical Research, Monroe, North Carolina
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee